CLINICAL TRIAL: NCT05015920
Title: A Phase 1 Open Label Study Evaluating the Safety and Efficacy of Gene Therapy in Subjects With β-Thalassemia Major by Transplantation of Autologous CD34+Stem Cells Transduced With a Lentiviral Vector Encoding βA-T87Q-Globin
Brief Title: A Study Evaluating the Safety and Efficacy of the BD211 Drug Product in β-Thalassemia Major Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai BDgene Co., Ltd. (Industry)
Collaborators: 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 920IEC/AF/61/2019-01.0
Record Dates: First submitted 2021-06-07; First posted 2021-08-23 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Hematologic Diseases
Keywords: TDT; β-thalassemia major
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobilization,harvest,transduction,conditioning,treatment,engraftment (Experimental): Subjects will participate in this study for a total of approximately 27 months, consisting of an up to 3 months pre-transplant period(consisting of a screening period followed by autologous cell harvest, followed by a waiting period during which the harvested cells are transduced and undergo release testing, followed by treatment with busulfan IV, and a single infusion of BD211 Drug Product) and a 24-month post-transplant evaluation period. Following completion of this study, all subjects will be asked to provided consent to participate in a follow-up study for another 13 years, which will focus on long-term safety, with an emphasis on integration site analysis, and long-term efficacy.
  Interventions: Genetic: BD211 Drug Product

INTERVENTIONS:
Genetic: BD211 Drug Product — Transplantation of Autologous CD34+Stem Cells Transduced to BD211 finished Product with a Lentiviral Vector coding βA-T87Q-Globin.

SUMMARY:
This is a Phase 1,open label,safety,and efficacy study in subjects with non-β0/β0 TDT β-thalassemia Major by transplanting BD211 drug product which is for autologous use only,via a single IV administration.

DETAILED DESCRIPTION:
After collection of mobilised peripheral blood samples, the patient's autologous cells,enriched for CD34+ HSCs, undergo ex vivo transduction with lentiviral vector encoding βA-T87Q-globin to BD211 finished product,which is then infused intravenously into the patient after myeloablative busulfan conditioning to prepare bone marrow "niches" for engraftment of the HSCs.

After discharge, subjects will be followed monthly, at a minimum, for 6 months and thereafter every 3 months for the remainder of the 24 months post-transplant.

Evaluation will include Routine and special biological testing at regular intervals, collection of AEs and concomitant medications, and evaluation of disease specific biological and clinical parameters.

Subjects will then be enrolled in a long-term follow-up protocol with annual evaluations for an additional 13 years post-transplant.

The long-term follow-up study will focus on long-term safety, with an emphasis on integration site analysis, and long-term efficacy.

This study will end when the last subject completes the Month 24 visit or discontinues from the study.

ELIGIBILITY:
Inclusion Criteria:

1. 5 to 35 years of age.
2. Be eligible for allogeneic HSCT based on institutional medical guideline, but without a matched related donor.
3. Transfusion-dependent β-Thalassemia Major, regardless of the genotype, with the diagnosis confirmed by Hb studies. Subjects must be stable and maintained on an appropriate iron chelation regimen. Transfusion dependence is defined as requiring at least 100 mL/kg/year of packed red blood cells(pRBCs).
4. Have been treated and followed for at least the past 2 years in a specialized center that maintained detailed medical records, including transfusion history.
5. Be willing and able, in the Investigator's opinion, to comply with the study procedures outlined in the study protocol. If a pediatric subject, the subject's parent/legal guardian also must be willing and able to comply with the study procedures outlined in the study protocol.

Exclusion Criteria:

1. Availability of a willing matched HLA-identical sibling hematopoietic cell donor.
2. Positive for presence of human immunodeficiency virus, human T-lymphotropic virus, vesicular stomatitis virus G antibody.
3. Clinically significant, active bacterial, viral, fungal, or parasitic infection.
4. A white blood cell (WBC) count<3x109/L and/or platelet count<120x109/L
5. Receipt of an allogeneic transplant.
6. Receipt of erythropoietin within 3 months before HSCT harvest.
7. Contraindication to anesthesia for bone marrow harvesting.
8. Any of prior or current malignancy, myeloproliferative or immunodeficiency disorder.
9. Active relapsing malaria
10. Immediate family member with a known or suspected Familial Cancer Syndrome.
11. Diagnosis of significant psychiatric disorder of the subject that could seriously impede the ability to participate in the study.
12. Pregnancy or breastfeeding in a postpartum female or absence of adequate contraception for fertile subjects.
13. Any other condition that would render the subject ineligible for HSCT, as determined by the attending transplant physician.
14. History of major organ damage.including Liver, Heart, Kidney disease, pulmonary hypertension ,severe iron overload, which in the opinion of the physician is grounds for exclusion.
15. Participation in another clinical study with an investigational drug within 30 days of screening.
16. Hydroxyurea therapy within 3 months before hematopoietic stem cell collection.
17. An assessment by the Investigator that the subject or parents of the subject will not comply with the study procedures outlined in the study protocol.
18. Subjects who have the desire to become a parent within the 27-month study period.
19. Prior receipt of gene therapy.

Ages: 5 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the success and kinetics of HSC engraftment. | At multiple timepoints after infusion for 24 months.
  Three consecutive absolute neutrophil counts≥500 cells/uL, three consecutive platelet values ≥20 e9/L, measure blood samples monthly after BD211 drug product infusion.
Incidence of transplant-related mortality through 100 days post-transplant. | Up to 100 days post-HSCT.
  Incidence of transplant-related mortality through 100 days post-transplant.
Overall survival of maintenance phase. | Up to 24 months post-HSCT.
  Overall survival up to 24 months post-HSCT.
Post-transplant blood samples for replication competent lentivirus (RCL) testing. | At multiple timepoints after infusion for 24 months.
  The testing of any subject positivity will be considered an SAE and suspend the inclusion of new subjects.
Assessment of Clonal dominance or leukemia/lymphoma and other malignancies. | At multiple timepoints after infusion for 24 months.
  Using peripheral blood of subjects for integration site analysis via LAM-PCR & deep sequencing.
Incidence of treatment- related adverse events. | Up to 24 months after BD211 drug product infusion.
  According to the requirements of the National Cancer Institute Common Terminology Standards for Adverse Events (NCI CTCAE) version 5.0, monitor laboratory parameters and the frequency and severity of clinical AEs.

SECONDARY OUTCOMES:
Quantify gene transfer efficiency and expression of BD211 drug product. | Up to 24 months after engraftment.
  Expression of βA-T87Q-globin chain in whole blood by assessing the ratio of βA-T87Q-globin to α-globin, as well as βA-T87Q-globin fractions in all β-chains over time by HPLC.
Quantify the hematopoietic chimerism resulting from treatment with BD211 drug product. | Up to 24 months after engraftment.
  Measuring lentiviral vector copy number per diploid genome(c/dg) for evaluation.
HbAT87Q in peripheral blood | Up to 24 months after engraftment.
  Measure the effects of transplantation with BD211 on the expression of disease-specific biological parameters and clinical events, including amounts of HbAT87Q in peripheral blood in grams per deciliter (g/dL).
Reduction of RBC transfusion requirements from baseline | Up to 24 months after engraftment.
  Reduction from baseline of RBC transfusion requirements (mL/kg) per month and year post-transplant, Up to 24 months after engraftment.
Duration of transfusion independence (months). | Up to 24 months after engraftment.
  Duration of transfusion independence up to 24 months after engraftment.
Weighted average Hemoglobin | Up to 24 months after engraftment.
  Weighted average Hemoglobin during transfusion independence in grams per deciliter (g/dL), up to 24 months after engraftment.
Changes of liver iron burden from baseline | Up to 24 months after engraftment.
  Changes from baseline in iron burden by assessing liver iron content (mg Fe/g dry weight).
Changes of cardiac iron burden from baseline | Up to 24 months after engraftment.
  Changes from baseline in iron burden by assessing cardiac iron content using magnetic resonance imaging (MRI) T2* value (milliseconds, ms).

CONTACTS AND LOCATIONS:
Overall Officials: Sanbin Wang, Dr., Study Chair — 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China
Locations (1):
- 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT05015920/ICF_000.pdf